CLINICAL TRIAL: NCT02532257
Title: An Open Label, Phase 2 Study of Ibrutinib in Combination With Rituximab and Lenalidomide in Previously Untreated Subjects With Follicular Lymphoma and Marginal Zone Lymphoma
Brief Title: Ibrutinib in Combination With Rituximab and Lenalidomide in Treating Patients With Previously Untreated, Stage II-IV Follicular Lymphoma or Marginal Zone Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0361; NCI-2015-01513 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0361 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Ann Arbor Stage II Follicular Lymphoma; Ann Arbor Stage II Marginal Zone Lymphoma; Ann Arbor Stage III Follicular Lymphoma; Ann Arbor Stage III Marginal Zone Lymphoma; Ann Arbor Stage IV Follicular Lymphoma; Ann Arbor Stage IV Marginal Zone Lymphoma; CD20 Positive; Grade 1 Follicular Lymphoma; Grade 2 Follicular Lymphoma; Grade 3a Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — ibrutinib; Lenalidomide; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lenalidomide, rituximab, ibrutinib) (Experimental): Patients receive lenalidomide PO on days 1-21, rituximab IV over 4-6 hours on days 1, 8, 15, and 22 of cycle 1 and day 1 of all subsequent cycles, and ibrutinib PO QD on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Biological: Rituximab

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima

SUMMARY:
This phase II trial studies how well ibrutinib in combination with rituximab and lenalidomide works in treating patients with previously untreated, stage II-IV follicular lymphoma or marginal zone lymphoma. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, may block cancer growth in different ways by targeting certain cells. Biological therapies, such as lenalidomide, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Giving ibrutinib in combination with rituximab and lenalidomide may work better in treating follicular lymphoma or marginal zone lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of ibrutinib combined with rituximab and lenalidomide in patients with previously untreated follicular lymphoma (FL) and marginal zone lymphoma (determined by progression-free survival at 2 years).

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of ibrutinib combined with rituximab and lenalidomide in subjects with FL as assessed by complete response rate (CR) at 120 weeks, overall response rate (ORR), duration of response (DOR), event free survival (EFS), time to next anti-lymphoma treatment (TTNT), and overall survival (OS).

II. To evaluate the safety and tolerability of ibrutinib combined with rituximab and lenalidomide in previously untreated subjects with FL and marginal zone lymphoma.

EXPLORATORY OBJECTIVES:

I. To evaluate prognostic and mechanistic biomarkers relative to treatment outcomes.

OUTLINE:

Patients receive lenalidomide orally (PO) on days 1-21, rituximab intravenously (IV) over 4-6 hours on days 1, 8, 15, and 22 of cycle 1 and day 1 of all subsequent cycles, and ibrutinib PO once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for 1 year and then every 24 weeks for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD20+ follicular lymphoma, grade 1, 2, or 3a or marginal zone lymphoma
* Have had no prior systemic treatment for lymphoma
* Bi-dimensionally measurable disease, with at least one mass lesion >= 2 cm in longest diameter by computed tomography (CT), positron emission tomography (PET)/CT, and/or magnetic resonance imaging (MRI)
* In the opinion of the investigator would benefit from systemic therapy
* Stage II, III, or IV disease
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count (ANC) >= 1,000/mm^3, independent of growth factor support (within 28 days prior to signing informed consent).
* Platelet counts >= 100,000/mm^3 or >= 50,000/mm^3 if bone marrow involvement with lymphoma, independent of transfusion support in either situation (within 28 days prior to signing informed consent).
* Serum aspartate transaminase (AST) or alanine transaminase (ALT) < 3 x upper limit of normal (ULN)
* Creatinine clearance > 30 ml/min calculated by modified Cockcroft-Gault formula
* Bilirubin < 1.5 x ULN unless bilirubin is due to Gilbert's syndrome, documented liver involvement with lymphoma, or of non-hepatic origin, in which case bilirubin should not exceed 3 g/dL
* Prothrombin time (PT)/international normalized ratio (INR) < 1.5 x ULN and partial thromboplastin time (PTT) < 1.5 x ULN
* Must be able to adhere to the study visit schedule and other protocol requirements
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study; females of childbearing potential: must either completely abstain from heterosexual sexual conduct or must use 2 methods of reliable contraception, 1 highly effective (intrauterine device, birth control pills, hormonal patches, injections, vaginal rings, or implants) and at least 1 additional method (condom, diaphragm, cervical cap) of birth control; reliable contraceptive methods must be started at least 4 weeks before lenalidomide; males who are sexually active must be practicing complete abstinence or agree to a condom during sexual contact with a pregnant female or female of child bearing potential; men must agree to not donate sperm during and after the study; for females, these restrictions apply at least 4 weeks before study treatment, during the period of therapy and for 1 month after the last dose of study drug; for males, these restrictions apply during the period of therapy and for 3 months after the last dose of study drug
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [Beta-hCG]) pregnancy test at screening; women who are pregnant or breastfeeding are ineligible for this study; females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid Risk Evaluation and Mitigation Strategy (REMS) program
* Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study
* All study participants must be registered into the mandatory Revlimid REMS program, and be willing and able to comply with the requirements of the REMS program

Exclusion Criteria:

* Known central nervous system lymphoma or leptomeningeal disease, except subjects with a history of central nervous system lymphoma treated and in remission > 6 months
* Evidence of diffuse large B-cell transformation
* Grade 3b FL
* Any prior history of other malignancy besides FL or marginal zone lymphoma, unless the patient has been free of disease for >= 5 years and felt to be at low risk for recurrence by the treating physician, except:

  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk, including but not limited to:

  * Moderate to severe hepatic impairment (Child-Pugh classes B and C)
* Known history of human immunodeficiency virus (HIV) or active hepatitis C virus or active hepatitis B virus infection, or any uncontrolled active systemic infection

  * Patients with inactive hepatitis B infection must adhere to hepatitis B reactivation prophylaxis unless contraindicated
* Prior use of ibrutinib or other BTK inhibitors, rituximab or lenalidomide
* Concurrent systemic immunosuppressant therapy (e.g., cyclosporine, tacrolimus, etc., or chronic administration glucocorticoid equivalent of > 10 mg/day of prednisone) within 28 days of the first dose of study drug
* Known anaphylaxis or immunoglobulin E (IgE)-mediated hypersensitivity to murine proteins or to any component of rituximab
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon); if patients have been on warfarin or equivalent vitamin K antagonists in the past, they will not be eligible if administered within 30 days of the first dose of study drug
* Requires chronic treatment with strong CYP3A inhibitors; if patients have been on a strong CYP3A inhibitor in the past, they will not be eligible if the CYP3A inhibitor was administered within 7 days of the first dose of study drug
* Requires chronic treatment with strong CYP3A inducers, for a list of strong CYP3A inducers, see the protocol. If patients have been on a strong CYP3A inducer in the past, they will not be eligible if the CYP3A inducer was administered within 7 days of the first dose of study drug
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association Functional classification
* Significant screening electrocardiogram (ECG) abnormalities including left bundle branch block, 2nd degree atrioventricular (AV) block, type II AV block, or 3rd degree block
* Known bleeding diathesis (e.g., von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 6 months prior to study entry
* Vaccinated with live, attenuated vaccines within 4 weeks of study entry
* Lactating or pregnant subjects
* Administration of any investigational agent within 28 days of first dose of study drug
* Patients who have undergone major surgery within 7 days or minor surgery within 3 days of first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loretta J Nastoupil, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Gordon MJ, Feng L, Strati P, Lee HJ, Hagemeister FB, Westin JR, Samaniego F, Marques-Piubelli ML, Vega Vazquez F, Parra Cuentas ER, Solis-Soto LM, Ma W, Wang J, Claret L, Averill B, Ibanez K, Fayad LE, Flowers CR, Green MR, Davis RE, Neelapu SS, Fowler NH, Nastoupil LJ. Safety and efficacy of ibrutinib in combination with rituximab and lenalidomide in previously untreated follicular and marginal zone lymphoma: An open label, phase 2 study. Cancer. 2024 Mar 15;130(6):876-885. doi: 10.1002/cncr.35114. Epub 2023 Nov 20. Erratum In: Cancer. 2025 Jun 15;131(12):e35933. doi: 10.1002/cncr.35933. PMID 37985359
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: 38 particpants previously untreated Follicular Lymphoma, 10 Marginal Zone Lymphoma
Period: Overall Study
Arm/Group | Arm 1
Started | 48
Previously Untreated Follicular Lymphoma FL Grade 1-3a | 38
Marginal Zone | 10
Completed | 29
Not Completed | 19
Not completed — Adverse Event | 2
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 3
Not completed — Progressive Disease | 10

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: 38 participants previously untreated Follicular Lymphoma, 10 Marginal Zone Lymphoma
Arm/Group | Arm 1
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 38
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Evaluate the efficacy of ibrutinib combined with rituximab and lenalidomide in patients with previously untreated FL and marginal zone lymphoma (determined by PFS at 2 years). Response will be assessed by the investigator based on the 2014 Cheson Lugano criteria. The 2-year PFS rate will be calculated and corresponding 95% confidence interval (CI) will be derived. Kaplan-Meier method will be used to estimate the PFS. Corresponding 95% CI will be summarized. Cox proportional hazards models will be used to assess the effects of patient prognostic factors on time-to-event endpoints.
Time Frame: 24 months
Population: 38 participants previously untreated Follicular Lymphoma, 10 Marginal Zone Lymphoma
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 48
percentage of participants
  PFS at 24 months (previously untreated Follicular Lymphoma): number analyzed (Participants) | 38
  PFS at 24 months (previously untreated Follicular Lymphoma) | 71.2 [57.7 to NA] — Not reached
  PFS at 24 months (mzl): number analyzed (Participants) | 10
  PFS at 24 months (mzl) | 54.2 [25.7 to NA] — Not reached

2. Secondary Outcome: Complete Response (CR) Rate
Description: Will be defined as the percentage of participants with a CR at 120 weeks as determined by the principal investigator (Cheson, Lugano classification 2014).
Time Frame: At 120 weeks
Population: 2 participants were unevaluable
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Arm 1
Number analyzed (Participants) | 46
percentage of participant | 63 [47.5 to 76.8]

3. Secondary Outcome: Overall Response Rate (ORR) (CR Rate + Partial Response [PR])
Description: Will be defined as the percentage of participants with an ORR and assessed by the investigator based on Cheson, Lugano 2014. The best ORR will be recorded.
Time Frame: Up to 3 years
Population: 2 participants were unevaluable
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 46
percentage of participants | 95.8 [85.7 to 99.5]

4. Secondary Outcome: Duration of Response (DOR)
Description: Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% CI.
Time Frame: Time by which measurement criteria for CR rate or PR, whichever is recorded first, is met until death or the first date by which progressive disease is documented; assessed up to 71.2 months
Population: 2 participants were unevaluable
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1
Number analyzed (Participants) | 46
months | 71.2 [57.7 to NA] — Not reached

5. Secondary Outcome: Event Free Survival (EFS)
Description: Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% CI.
Time Frame: From the date of course 1, day 1 to the date of first documented progression, transformation to diffuse large B-cell lymphoma, initiation of new anti-lymphoma treatment, or death; assessed up to 70.2 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1
Number analyzed (Participants) | 48
months | 70.2 [53.4 to NA] — Not reached

6. Secondary Outcome: Time to Next Anti-lymphoma Treatment (TTNT)
Description: Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% CI.
Time Frame: From the date of course 1, day 1 to the date of first documented administration of any anti-lymphoma treatment (chemotherapy, radiotherapy, immune therapy, radioimmunotherapy, or other experimental therapy); assessed up to 75.8 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1
Number analyzed (Participants) | 48
months | 75.8 [70.5 to NA] — Not reached

7. Secondary Outcome: Overall Survival (OS) Rate
Description: Secondary endpoints included best and 120 week complete response rate (CRR) and ORR by Lugano classification, duration of response, event free survival, time to next anti-lymphoma treatment, overall survival (OS) and safety. Response evaluation was performed at cycle 4, day 1, cycle 7 day 1, at the end of cycle 12, then every 12 weeks for the first four assessments, then every 24 weeks until disease progression
Time Frame: From the date of course 1, day 1 to the date of death regardless of cause; assessed up to 78 months
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 48
percentage of participants | 97.9

ADVERSE EVENTS:
Time Frame: 4 years, 1 month
Description: The time a subject has signed and dated an Informed Consent Form (ICF) until completion of the subject's last study-related procedure (which may include contact for follow-up safety).
Arm/Group | Arm 1
All-Cause Mortality (participants affected / at risk) | 1/48
Serious Adverse Events (participants affected / at risk) | 24/48
Other Adverse Events (participants affected / at risk) | 40/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=48)
Diarrhea (Gastrointestinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (Nervous system disorders) | 2
Pruritis (Skin and subcutaneous tissue disorders) | 1
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 24
Anemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=48)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Blurred Vision (Eye disorders) | 5
Chills (Infections and infestations) | 15
Constipation (Gastrointestinal disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 23
Edema, limbs (Blood and lymphatic system disorders) | 18
Fatigue (Nervous system disorders) | 35
Fever (Infections and infestations) | 11
Headache (General disorders) | 17
Mucositis (Gastrointestinal disorders) | 12
Myalgia (Nervous system disorders) | 37
Nausea (Gastrointestinal disorders) | 16
Numbness (Nervous system disorders) | 7
Pruritis (Skin and subcutaneous tissue disorders) | 7
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 16
Vomiting (Gastrointestinal disorders) | 5
Anemia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 0
Neutropenia (Blood and lymphatic system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT02532257/Prot_SAP_000.pdf